CLINICAL TRIAL: NCT01528202
Title: Effect of Tart Cherry Juice (Prunus Cerasus) on Melatonin Levels and Sleep Quality
Brief Title: Tart Cherries and Melatonin Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: University of Surrey (Other)
Responsible Party: Principal Investigator, Dr. Glyn Howatson, Laboratory Director, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SLS_SUB60
Record Dates: First submitted 2012-02-03; First posted 2012-02-07 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Sleep
Keywords: Sleep, circadian cycle, melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Baseline placebo (No Intervention): measures taken before administration of placebo
- Placebo (Placebo Comparator): Placebo intervention given after 'baseline placebo' arm
  Interventions: Dietary Supplement: Fruit juice cordial
- baseline cherry juice (No Intervention): measures taken before the cherry juice intervention
- cherry juice (Experimental): trial where cherry juice is taken following the 'baseline cherry juice' arm
  Interventions: Dietary Supplement: Cherry juice

INTERVENTIONS:
Dietary Supplement: Cherry juice — 30 mLs preceding morning meal and 30 mLs preceding evening meal each day for 7 days.
  Other Names: CherryActive concentrate
  Arms: cherry juice
Dietary Supplement: Fruit juice cordial — fruit flavoured juice concentrate
  Other Names: Apple and blackcurrent squash (0164 9338). Sainsbry's Supermarkets Ltd.
  Arms: Placebo

SUMMARY:
The aim of this investigation was to examine the effects of tart Montmorency cherry juice on urinary 6-sulfatoxymelatonin and sleep quality using a double-blind, placebo-controlled, cross-over design.

DETAILED DESCRIPTION:
The aim of the study is to examine the efficacy of tart cherry juice on sleep quality, quantity, and timing. Naturally circulating melatonin is instrumental in regulating sleep/wake schedules. Tart Montmorency cherries (Prunus Cerasus) contain high levels of melatonin and may be a useful intervention to supplement for realignment of circadian phase and by increasing the robustness of circadian amplitude. In normal healthy adults, with experimentally induced phase advanced circadian misalignment, the administration of a 3mg supplement of melatonin significantly increased sleep architecture characteristics. In this study we want to examine the efficacy of tart cherry juice in increasing urinary levels of melatonin and the subsequent impact this will have on sleep parameters.

ELIGIBILITY:
Inclusion Criteria:

* Equal numbers of healthy, non-pathological males and females aged between 18-39.

Exclusion Criteria:

* history of epilepsy, current episode of major depressive disorder or anxiety disorder, or a current sleep problem or an inability to comprehend English, travel over two time zones within the last six months, excessive alcohol (over 3 units per day) or caffeine consumption (more than 6 caffeinated drinks or 1 after 6pm), a smoker, a shift worker, a familial history of diabetes, users of medication or supplements, or if the participant is pregnant or currently lactating.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
urinary 6-sulphatoxymelatonin | continually for 48 hours
  urinary 6-sulphatoxymelatonin is the primary metabolite of melatonin and provides a sarrogate marker of melatonin metabolism. By measuring over a 48 h period it is possible to examine the circadian rhythm of melatonin.

SECONDARY OUTCOMES:
Sleep quality | continually throughout the duration of the study
  Acti watches quantitively measure sleep and activity of participants, whereas slep recall provides a retrospective and subjective m,easure of sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom